CLINICAL TRIAL: NCT05919979
Title: Efecto de Una sesión de Ejercicio físico Realizada Durante un Periodo de Ayuno de 24-34 Horas Sobre el Metabolismo energético y la función Cognitiva en Adultos Sanos: Estudio Piloto
Brief Title: Effect of a Physical Exercise Session Performed During a 24-34 Hour Fasting Period on Energy Metabolism and Cognitive Function in Healthy Adults
Acronym: IMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: University Hospital Virgen de las Nieves (Other)
Responsible Party: Principal Investigator, Guillermo Sanchez Delgado, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GSD-2023-002
Record Dates: First submitted 2023-06-05; First posted 2023-06-27 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Energy Metabolism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting, then fasting+exercise (Experimental)
  Interventions: Behavioral: 34-hour fasting in sedentary conditions; Behavioral: 34-hour fasting with high-intensity exercise
- Fasting + Exercise, then fasting (Experimental)
  Interventions: Behavioral: 34-hour fasting in sedentary conditions; Behavioral: 34-hour fasting with high-intensity exercise

INTERVENTIONS:
Behavioral: 34-hour fasting in sedentary conditions — Participants will fast for 34h after a standardized breakfast, refraining from physical activity.
Behavioral: 34-hour fasting with high-intensity exercise — Participants will fast for 34h after a standardized breakfast, performing a high-intensity exercise session 6-10 hours aprox. after starting the fasting period.

SUMMARY:
This study explores the impact of high-intensity exercise during fasting on energy metabolism and cognitive function in healthy adults. Changes in respiratory exchange ratio, blood substances, and cognitive performance will be measured after 24 and 34 hours of fasting with and without exercise in a randomized crossover design.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years old.
* Body mass index: 18.5-30.0 Kg/m2.
* Stable body weight (5kg range within the last 3 months)
* Being able to consume all the food items provided as part of the study.
* Not having change the time zone or have shifted sleeping hours equivalent to more than 3 hours on the previous 2 weeks.

Exclusion Criteria:

* Diagnosed with any chronic condition that, in the research team's opinion or based on the American College of Sports Medicine guidelines, could contraindicate the implementation of 34-hour fasting periods and/or high-intensity exercise.
* Diagnosed with a chronic endocrine, digestive, rheumatic, neurological, cardiac, pulmonary, autoimmune, or infectious condition that affects energy metabolism.
* Presenting any signs or symptoms of illness that, in the research team's opinion or based on the American College of Sports Medicine guidelines, could contraindicate the implementation of 34-hour fasting periods and/or high-intensity exercise.
* Pregnant or breastfeeding.
* Using medications or supplements that may alter energy metabolism.
* Currently undergoing or having undergone any type of nutritional intervention or treatment in the past 3 months.
* Engaging in more than 5 hours per week of habitual moderate-to-vigorous cycling.
* Any other condition that, in the research team's opinion, discourages participation in the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2023-05-29 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Respiratory Exchange Ratio | 24-hour after starting the fasting period

SECONDARY OUTCOMES:
Respiratory Exchange Ratio | 34-hour after starting the fasting period
Serum insulin concentration | 24-hour after starting the fasting period
Serum insulin concentration | 34-hour after starting the fasting period
Serum glucose concentration | 24-hour after starting the fasting period
Serum glucose concentration | 34-hour after starting the fasting period
Dimensional Change Card Sort Test (NIH toolbox) | 24-hour after starting the fasting period
Dimensional Change Card Sort Test (NIH toolbox) | 34-hour after starting the fasting period
List Sorting Working Memory Test (NIH toolbox) | 24-hour after starting the fasting period
List Sorting Working Memory Test (NIH toolbox) | 34-hour after starting the fasting period
Flanker Test (NIH toolbox) | 24-hour after starting the fasting period
Flanker Test (NIH toolbox) | 34-hour after starting the fasting period

CONTACTS AND LOCATIONS:
Locations (1):
- Instiuto Mixto Universitario Deporte y Salud, Granada, Granada, Spain